CLINICAL TRIAL: NCT05319470
Title: Ocular Surface Disease and IOP Monitoring With Travoprost Without Conservatives
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES3/Th11/03-02-2022
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma; Glaucoma; Drugs; Ocular Surface Disease
Keywords: glaucoma; travoprost; prostaglandin without preservatives
MeSH Terms: conditions — Glaucoma | interventions — Intraocular Pressure; Wettability; Visual Fields

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: 100 patients with diagnosed glaucoma receiving travoprost without preservatives
  Interventions: Diagnostic Test: Intraocular pressure (IOP); Diagnostic Test: Tear Break-up Time (TBUT); Diagnostic Test: Conjuctival Hyperemia; Diagnostic Test: Schirmer Test; Diagnostic Test: Visual Fields and OCT RNFL

INTERVENTIONS:
Diagnostic Test: Intraocular pressure (IOP) — Measurement of intraocular pressure in both eyes of the study population using the Goldman applanation tonometer.
Diagnostic Test: Tear Break-up Time (TBUT) — TBUT will be calculated after instillation of a drop of fluorescein dye, by slit lamp biomicroscopy.
Diagnostic Test: Conjuctival Hyperemia — Conjunctival hyperemia will be assessed by slit lamp biomicroscopy using a validated grading system.
Diagnostic Test: Schirmer Test — Schirmer test will be performed on both eyes to asses tear production.
Diagnostic Test: Visual Fields and OCT RNFL — Visual field examination using a Humphrey perimeter and measurement of peripapillary retinal nerve fiber layer thickness with optical coherence tomography.

SUMMARY:
Primary objective of this study is to study the efficacy of travoprost without preservatives in the treatment of glaucoma patients and to monitor the ocular surface.

DETAILED DESCRIPTION:
This is a prospective study including patients visiting the outpatient glaucoma clinic of the University General Hospital of Alexandroupolis for their standard evaluation. Study population is already under treatment with a travoprost preparation without preservatives. They will be fully informed about the procedure and the purpose of the study and a written consent will be obtained. For every patient included in the study intraocular pressure will be measured using a Goldman applanation tonometer, according to the standard way of practice at our clinic. Also, Tear Break-Up-Time (BUT), conjunctival hyperemia grading and Schirmer testing will be used to assess the ocular surface state. Visual field tests and OCT RNFL measurements will also be obtained. The above measurements will be repeated 6 months after the initial examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma treated with travoprost without preservatives.

Exclusion Criteria:

* Co-administration of another anti-glaucoma preparation with or without preservatives, Sjogren's syndrome, poor eyelid occlusion of any etiology.

Ages: 35 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult glaucoma patients already under treatment with travoprost without preservatives.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | 6 months
  Intraocular pressure measurement in both eyes using the Goldman applanation tonometer.
Ocular Surface Disease | 6 months
  Tear breakup time (TBUT), conjuctival hyperemia scoring and Schirmer testing will be used to assess the ocular surface state of the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD,PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: Undecided